CLINICAL TRIAL: NCT00521118
Title: A Phase II Study to Determine the Response to Second Curettage as Initial Management for Persistent Low Risk, Non-metastatic Gestational Trophoblastic Neoplasia
Brief Title: Second Curettage in Treating Patients With Persistent Non-metastatic Gestational Trophoblastic Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0242; NCI-2009-00606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0242; CDR0000561984; GOG-0242 (Other: NRG Oncology); GOG-0242 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Complete Hydatidiform Mole; Non-Metastatic Gestational Trophoblastic Tumor; Partial Hydatidiform Mole
MeSH Terms: conditions — Hydatidiform Mole

ARMS (1):
- Treatment (second curettage) (Experimental): Patients undergo a second curettage rather than standard treatment (immediate chemotherapy) within 14 days of registration.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo second curettage

SUMMARY:
This phase II trial studies how well a second curettage (removal of the abnormal cancer cells in the uterus using a method of surgically removing the lining of the uterus) works in treating patients with gestational trophoblastic tumors that did not go away after a first curettage (persistent) and has not yet spread to other places in the body (non-metastatic). A second curettage may be effective in treating persistent gestational trophoblastic tumors and may decrease the likelihood that patients will need chemotherapy in the near future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response to second curettage in patients with persistent, non-metastatic gestational trophoblastic neoplasia (GTN).

SECONDARY OBJECTIVES:

I. To evaluate if response to a second curettage is independent of the tumor burden as measured by the quantitative beta-human chorionic gonadotropin (hCG) assay at study entry.

II. To evaluate if response to a second curettage is independent of the depth of myometrial invasion as measured sonographically following the initial curettage but prior to study entry (when persistent disease is first diagnosed).

III. To estimate the frequency of complications related to a second curettage, specifically infection of the fallopian tubes or ovaries, hemorrhage associated with curettage, or operative injury to the uterus.

IV. To estimate the frequency of a change in the uterine histology between the first and second curettage.

OUTLINE:

Patients undergo a second curettage rather than standard treatment (immediate chemotherapy) within 14 days of registration.

After completion of study treatment, patients are followed up at 14 days, weekly for 4 weeks, and then monthly for 5 months, and then every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had hydatidiform mole treated by evacuation and/or curettage and now meet the criteria of low risk GTN, as defined by the International Federation of Gynecology and Obstetrics (F.I.G.O.)/World Health Organization (W.H.O.) 2002 staging and risk scoring criteria:

  * A plateau in the beta-hCG assay for 4 consecutive weekly levels over a period of 3 weeks or longer; that is, days 1, 7, 14, 21; for this study, a plateau will be defined as less than a 10% decline using as a reference the initial value in the series of values taken over a period of 3 weeks; OR
  * A rise in the beta-hCG assay of 3 consecutive measurements, or longer, over at least a period of 2 weeks or more; days, 1, 7, 14; for this study, a rise will be defined as an increase of greater than 20% taking as a reference the initial value in the series of values taken over the 2-week period; OR
  * When the beta-hCG level remains elevated above normal for 6 months or longer
* Patients must have a clinically significant elevated beta-hCG level of greater than 20 mIU/ml
* Patients must have non-metastatic low risk GTN with a W.H.O. 2002 risk score of no greater than 6
* Patients must have no metastatic disease as determined by the pelvic examination, pelvic ultrasound, and chest x-ray
* Patients must have signed an approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0 or 1
* Patients must have histologically confirmed complete or partial mole
* Patients must agree to use an accepted method of contraception (oral contraceptives, birth control patches, Depo-Provera, diaphragm, contraceptive foam and condom, or male/female sterilization)
* Patients must meet pre-entry requirements

Exclusion Criteria:

* Patients who do not have persistent low-risk GTN
* Patients with any evidence of metastatic disease beyond the uterus
* Patients with persistent or recurrent GTN (same gestation) that have already been treated with chemotherapy
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, patients who have had any evidence of the other cancer present within the last 5 years or patients whose previous cancer treatment contraindicates this protocol therapy
* Patients with histologically confirmed choriocarcinoma, placental site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT) on the first curettage
* Patients who refuse to use an accepted method of contraception
* Patients who have had more than one curettage for the management of the current disease or who have undergone hysterectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10-09 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2015-06-25 (Actual)

PRIMARY OUTCOMES:
Development of "second persistent" disease, defined as failure to achieve or maintain a normal assay, or a plateau, or a rise in the assay level after second curettage | Up to 6 months
Frequency of surgical cure defined as normal beta-hCG level documented for 6 consecutive months AND no chemotherapy | Up to 6 months
Incidence of adverse effects of second curettage, assessed by Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after the surgical procedure
  The frequency and severity of the reported adverse effects of repeat evacuation will be tabulated. Specifically, uterine operative injury, hemorrhage, and infection (pelvis, fallopian tubes and ovaries) will be prospectively collected.
Surgical failure, defined as the development of choriocarcinoma, placental site trophoblastic tumor, or epithelioid trophoblastic tumor histologically diagnosed at second curettage | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Osborne, Principal Investigator — NRG Oncology
Locations (29):
- United States (28):
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Memorial University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Gynecologic Oncology Network, Greenville, North Carolina
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Osborne RJ, Filiaci VL, Schink JC, Mannel RS, Behbakht K, Hoffman JS, Spirtos NM, Chan JK, Tidy JA, Miller DS. Second Curettage for Low-Risk Nonmetastatic Gestational Trophoblastic Neoplasia. Obstet Gynecol. 2016 Sep;128(3):535-542. doi: 10.1097/AOG.0000000000001554. PMID 27500329